CLINICAL TRIAL: NCT00112840
Title: A Phase I/II Trial of CCI-779 and Bevacizumab in Stage IV Renal Cell Carcinoma
Brief Title: CCI-779 and Bevacizumab in Treating Patients With Metastatic or Unresectable Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00109; NCI-2009-00109 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000428311; NCI-6986; MC0452 (Other: Mayo Clinic); 6986 (Other: CTEP); N01CM62205 (NIH)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — temsirolimus; Bevacizumab

ARMS (1):
- CCI-779 and bevacizumab (Experimental): Patients receive CCI-779 IV on days 1, 8, 15, and 22 and bevacizumab IV on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of CCI-779 and bevacizumab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Phase II patients receive CCI-779 and bevacizumab as in phase I at the MTD determined in phase I. After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 3 years after study entry.
  Interventions: Drug: CCI-779; Drug: Bevacizumab

INTERVENTIONS:
Drug: CCI-779 — CCI-779 is taken IV on days 1, 8, 15, 22 of a 28-day cycle. Dose level is dependent on phase.
  Other Names: Temsirolimus; Torisel Rapamycin analog; WAY-130779
Drug: Bevacizumab — Bevacizumab is taken IV on Days 1 and 15 of a 28-day cycle. Dose Level determined by phase.

SUMMARY:
This phase I/II trial is studying the side effects and best dose of CCI-779 and bevacizumab and to see how well they work in treating patients with metastatic or unresectable kidney cancer. Drugs used in chemotherapy, such as CCI-779, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of kidney cancer by blocking blood flow to the tumor. Giving CCI-779 together with bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose (MTD) and recommended dosing for the combination of CCI-779 and Bevacizumab in patients with metastatic renal cell cancer. (Phase I) II. To determine the proportion of patients with metastatic renal cell cancer who are progression free at 6 months. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the toxicity of the combination of CCI 779 and Bevacizumab in patients with metastatic renal cell cancer. (Phase II) II. To determine the clinical response rate of CCI 779 and Bevacizumab in patients with metastatic renal cell cancer. (Phase II) III. To determine the time to progression (TTP), disease free survival, and overall survival of CCI 779 and Bevacizumab in patients with metastatic renal cell cancer. (Phase II)

TERTIARY OBJECTIVES:

I. To identify predictive molecular markers of response, both at the tumor level and in the plasma/serum level, in an exploratory manner.

II. To correlate blood markers of angiogenesis with clinical activity of the combination of CCI-779 and Bevacizumab.

OUTLINE: This is a multicenter, phase I dose-escalation study followed by a phase II study. Patients are stratified according to study phase (I vs II).

Phase I: Patients receive CCI-779 IV on days 1, 8, 15, and 22 and bevacizumab IV on days 1 and 15.

Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of CCI-779 and bevacizumab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Phase II: Patients receive CCI-779 and bevacizumab as in phase I at the MTD determined in phase I. After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 3 years after study entry.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or unresectable renal cell cancer

  * Must have a component of conventional clear cell histology
  * The following histologies are excluded:

    * True papillary
    * Sarcomatoid features without any clear cell component
    * Chromophobe
    * Oncocytoma
    * Collecting duct tumors
    * Transitional cell carcinoma
* Measurable disease, defined as ≥ 1 lesion ≥ 2.0 cm in the longest diameter by conventional techniques OR ≥ 1.0 cm by spiral CT scan
* Tumor tissue (from primary tumor or metastases) available AND patient is willing to donate blood for research studies (phase II only)
* No CNS metastases by head CT scan or MRI
* Performance status - ECOG 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* No evidence of bleeding diathesis or coagulopathy
* No history of clinically significant bleeding or active bleeding
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN (5 times ULN if liver metastases are present)
* AST ≤ 2.5 times ULN (5 times ULN if liver metastases are present)
* PT/INR ≤ 1.5

  * Patients on full-dose warfarin or stable-dose low molecular weight heparin must have INR > 1.5 but ≤ 3
* Creatinine ≤ 1.5 times ULN
* Urine protein ≤ 1+ by dipstick or urinalysis
* Urine protein < 1,000 mg on a 24-hour urine collection
* No cerebrovascular accident within the past 6 months
* No peripheral vascular disease with claudication on < 1 block
* No New York Heart Association class II-IV congestive heart failure
* No angina pectoris requiring nitrate therapy
* No myocardial infarction within the past 6 months
* No uncontrolled hypertension, defined as systolic blood pressure (BP) ≥ 160 mm Hg and/or diastolic BP ≥ 90 mm Hg despite medication
* No cardiac arrhythmias
* No other significant cardiovascular disease
* No ongoing hemoptysis
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3-4 months after study participation
* Fasting cholesterol ≤ 350 mg/dL
* Triglycerides ≤ 1.5 times ULN (may achieve using lipid lowering agents)
* No known hypersensitivity to recombinant human antibodies
* No significant traumatic injury within the past 4 weeks
* No serious or non-healing wound, ulcer, or bone fracture
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 4 weeks
* No pathological conditions that confer a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* No diabetes
* No other currently active malignancy except nonmelanoma skin cancer

  * Patients are not considered to have a currently active malignancy if they have completed anticancer therapy AND are considered to be at < 30% risk of relapse
* No other uncontrolled serious medical or psychiatric condition
* At least 4 weeks since prior biologic response modifiers for metastatic disease
* No prior bevacizumab or mTOR inhibitors
* At least 4 weeks since prior chemotherapy for metastatic disease
* Prior palliative radiotherapy to metastatic lesions allowed provided there is ≥ 1 measurable and/or evaluable lesion that has not been irradiated
* At least 4 weeks since prior and no concurrent radiotherapy
* Prior nephrectomy allowed
* More than 4 weeks since prior major surgery or open biopsy
* More than 1 week since prior core biopsy
* No concurrent major surgery
* At least 4 weeks (2 weeks for vascular endothelial growth factor [VEGF] receptor tyrosine kinase inhibitor [RTKI] therapy) since prior and no more than 2 therapies (phase II)

  * One of these therapies must have included a RTKI agent administered for a minimum of 4 weeks
* Concurrent full-dose warfarin or low molecular weight heparin allowed provided dose is stable AND INR requirements are met
* Concurrent zoledronate for bone metastases and/or hypercalcemia allowed provided therapy was initiated prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-05; Primary Completion 2010-08-09 (Actual); Study Completion 2015-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Merchan, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 5/11/2005 to 7/19/2006, 14 participants were registered to the Phase I portion of the study (8 at Dose Level 1 and 6 at Dose Level 2). Phase II opened 02/09/2007 at Dose Level 2 and registered 46 patients before closing with full accrual on 6/15/2010.
Pre-assignment Details: In Phase I, Dose Level 2, 2 subjects were unevaluable because they were removed from the study before completing cycle 1 of treatment for reasons other than toxicity. In Phase II, 5/46 patients were ineligible and one patient cancelled.
Groups:
- Phase I, Dose Level 1: Patients receive CCI-779 IV on days 1, 8, 15, and 22 and bevacizumab IV on days 1 and 15 In the Phase 1, Dose Level 1 portion, cohorts of 3-6 eligible patients were treated with CCI-779 (25 mg IV weekly) and IV Bevacizumab (level 1=5mg/kg) every other week. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase I, Dose Level 2: Patients receive CCI-779 IV on days 1, 8, 15, and 22 and bevacizumab IV on days 1 and 15 In the Phase 1, Dose Level 2 portion, cohorts of 3-6 eligible patients were treated with CCI-779 (25 mg IV weekly) and IV Bevacizumab (level 1= 10 mg/kg) every other week. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase II: Phase II patients were treated at the highest dose level (dose level 2: CCI-779 25 mg IV weekly and Bevacizumab 10 mg/kg IV every two weeks). Patients receive 25 mg CCI-779 IV on days 1, 8, 15, and 22 and 10 mg/kg bevacizumab IV on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 3 years after study entry.
Period: Overall Study
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase II
Started | 8 | 6 | 46
Completed | 6 | 6 | 40
Not Completed | 2 | 0 | 6
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Phase I, Dose Level 2: Patients receive CCI-779 IV on days 1, 8, 15, and 22 and bevacizumab IV on days 1 and 15 In the Phase 1, Dose Level 2 portion, cohorts of 3-6 eligible patients were treated with CCI-779 (25 mg IV weekly) and IV Bevacizumab (level 1=5mg/kg) every other week. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase II | Total
Number analyzed (Participants) | 8 | 6 | 46 | 60
Age, Continuous [Median (Full Range); unit: years] | 61 [44 to 75] | 66 [61 to 77] | 62 [38 to 82] | 62.5 [38 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 11 | 13
  Male | 7 | 5 | 35 | 47
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 46 | 60

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity (DLT) (Phase I)
Description: For this protocol, dose limiting toxicity (DLT) will be defined as an adverse event attributed (definitely, probably, or possibly) to the study treatment in the first four weeks of combination therapy, and meeting the following criteria:
  * Grade 4 Absolute neutrophil count (ANC) for 5+ days.
  * Grade 4 anemia or thrombocytopenia of any duration.
  * Serum Creatinine 2 times baseline or 2x upper limit of normal if baseline levels not normal.
  * Any other non-hematologic grade 3 or higher as per NCI Common Terminology Criteria for Adverse Events (CTCAE) v. 3.0, except fatigue and grade 3 Hypertension that is will be controlled with oral medication.
  * Grade 3 triglycerides will be a DLT for patients who have Grade 3 in spite of appropriate lipid lowering drug therapy.
  The maximum tolerated dose level (MTD) will be defined as the highest safely tolerated dose where 1 or 0 out of 6 patients experience DLT with the next higher dose.
Time Frame: Patients observed a minimum of 4 weeks (one full course). The maximum number of cycles observed was 16 cycles.
Measure: Number; unit: participants
Groups:
- Phase I, Dose Level 1: Patients receive CCI-779 IV on days 1, 8, 15, and 22 and bevacizumab IV on days 1 and 15 in escalating dose levels to determine Maximum Tolerated Dose (MTD). In the phase I portion, cohorts of 3-6 eligible patients were treated with CCI-779 (25 mg IV weekly) and doses of IV Bevacizumab (level 1=5mg/kg; level 2=10 mg/kg) every other week. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. The first three patients began at dose level 1 and cohort doses escalate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 3 years after study entry.
- Phase 1 , Dose Level 2: Patients receive CCI-779 IV on days 1, 8, 15, and 22 and bevacizumab IV on days 1 and 15 In the Phase 1, Dose Level 2 portion, cohorts of 3-6 eligible patients were treated with CCI-779 (25 mg IV weekly) and IV Bevacizumab (level 1=10 mg/kg) every other week. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Phase I, Dose Level 1 | Phase 1 , Dose Level 2 | Phase II
Number analyzed (Participants) | 6 | 6 | 0
participants | 1 | 1 |

2. Primary Outcome: Proportion of Progression-free Patients at 6 Months (Phase II)
Description: Determination of progression will be made according to Response Evaluation Criteria in Solid Tumors (RECIST). A progression (PD) is defined as having at least a 20% increase in the sum of the longest dimension of target lesions taking as reference the smallest sum of the largest dimension recorded at baseline.The proportion of progression-free patients will be estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the success proportion will be calculated. All patients meeting the eligibility criteria who have signed a consent form and begun treatment will be considered evaluable. Those who die will be considered to have had disease progression unless documented evidence clearly indicates no progression has occurred.
Time Frame: 6 months after study entry
Population: Only Phase II participants were analyzed for this endpoint. Forty participants from Phase II were evaluable for this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase I, Dose Level 1: Patients receive CCI-779 IV on days 1, 8, 15, and 22 and bevacizumab IV on days 1 and 15 in escalating dose levels to determine Maximum Tolerated Dose (MTD). In the phase I portion, cohorts of 3-6 eligible patients were treated with CCI-779 (25 mg IV weekly) and escalating doses of IV Bevacizumab (level 1=5mg/kg; level 2=10 mg/kg) every other week. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. The first three patients began at dose level 1 and cohort doses escalate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 3 years after study entry.
- Phase 1, Dose Level 2: Patients receive CCI-779 IV on days 1, 8, 15, and 22 and bevacizumab IV on days 1 and 15 In the Phase 1, Dose Level 2 portion, cohorts of 3-6 eligible patients were treated with CCI-779 (25 mg IV weekly) and IV Bevacizumab (level 1=10 mg/kg) every other week. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Phase I, Dose Level 1 | Phase 1, Dose Level 2 | Phase II
Number analyzed (Participants) | 0 | 0 | 40
percentage of participants |  |  | 40 [25 to 55]

3. Secondary Outcome: Clinical Best Response Rate of CCI-779 and Bevacizumab in Patients With Metastatic Renal Cell (Phase II)
Description: The number of participants with clinical tumor response to treatment will be evaluated using the Response Evaluation Criteria In Solid Tumors (RECIST).
  Complete Response (CR): Disappearance of all target lesions
  Partial Response (PR): At least a 30% decrease in the sum of the largest dimension (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: Up to 3 years from study registration
Population: All eligible Phase II patients were used to assess this endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 40
percentage of participants
  Partial Response (PR) | 20
  Complete Response (CR) | 0

4. Secondary Outcome: Time to Progression (Phase II)
Description: The time to progression is defined as the time from registration to the time of progression. Those who die will be considered to have had disease progression unless documented evidence clearly indicates no progression has occurred. The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years from study registration
Population: All eligible participants in Phase II were used for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 40
months | 7.6 [4.0 to 7.8]

5. Secondary Outcome: Overall Survival (Phase I and II)
Description: The overall survival or survival time is defined as the time from registration to death due to any cause. The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years from study registration
Population: All eligible participants were used for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 1, Dose Level 1: Patients receive CCI-779 IV on days 1, 8, 15, and 22 and bevacizumab IV on days 1 and 15 in escalating dose levels to determine Maximum Tolerated Dose (MTD). In the phase I portion, cohorts of 3-6 eligible patients were treated with CCI-779 (25 mg IV weekly) and doses of IV Bevacizumab (level 1=5mg/kg; level 2=10 mg/kg) every other week. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. The first three patients began at dose level 1 and cohort doses escalate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 3 years after study entry.
- Phase I, Dose Level 2: Patients receive CCI-779 IV on days 1, 8, 15, and 22 and bevacizumab IV on days 1 and 15 In the Phase 1, Dose Level 2 portion, cohorts of 3-6 eligible patients were treated with CCI-779 (25 mg IV weekly) and IV Bevacizumab (level 1=10 mg/kg) every other week. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Phase 1, Dose Level 1 | Phase I, Dose Level 2 | Phase II
Number analyzed (Participants) | 6 | 6 | 40
months | 24.4 [4.6 to NA] — Upper 95% confidence limit wasn't calculable due to an insufficient number of events | 17 [4.4 to 54.8] | 20.6 [11.5 to 23.7]

ADVERSE EVENTS:
Description: All patients that began study treatment and were assessed for adverse events are included in this report. Of the 46 patients that registered, one patient canceled prior to treatment and was not assessed for adverse events. Therefore, 45 patients are used in this report.
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase II
Serious Adverse Events (participants affected / at risk) | 3/8 | 2/6 | 12/45
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Dose Level 1 (N=8) | Phase I, Dose Level 2 (N=6) | Phase II (N=45)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 2 (2)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Peritoneal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Dose Level 1 (N=8) | Phase I, Dose Level 2 (N=6) | Phase II (N=45)
Hemoglobin decreased (Blood and lymphatic system disorders) | 7 (23) | 6 (25) | 40 (161)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac pain (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 0 (0) | 0 (0) | 1 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 1 (3) | 4 (5)
Anal exam abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 3 (13) | 5 (13) | 18 (54)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 1 (2) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 1 (2) | 7 (9)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (10) | 4 (9) | 26 (73)
Nausea (Gastrointestinal disorders) | 2 (3) | 3 (5) | 10 (21)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (4)
Proctitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Proctoscopy abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Tooth development disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (5)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (4) | 3 (5)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Chills (General disorders) | 1 (1) | 0 (0) | 3 (6)
Edema limbs (General disorders) | 0 (0) | 1 (3) | 5 (7)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 2 (6) | 5 (23) | 35 (171)
Fever (General disorders) | 0 (0) | 1 (1) | 4 (5)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 5 (7)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 3 (3)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 7 (16)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (7) | 10 (24)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 11 (25)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Creatinine increased (Investigations) | 5 (22) | 3 (7) | 26 (145)
INR increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 0 (0) | 1 (1) | 3 (10)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (9) | 2 (3) | 1 (2)
Neutrophil count decreased (Investigations) | 3 (5) | 3 (5) | 3 (6)
Platelet count decreased (Investigations) | 3 (7) | 4 (16) | 19 (57)
Serum cholesterol increased (Investigations) | 3 (25) | 6 (20) | 31 (115)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (9) | 10 (29)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (4) | 5 (23) | 18 (47)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 14 (56)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (6)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (18)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2) | 4 (7) | 11 (20)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 4 (7)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 3 (8) | 1 (2) | 10 (14)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 3 (6)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (5)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (13)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum triglycerides increased (Metabolism and nutrition disorders) | 3 (14) | 3 (16) | 33 (132)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (8)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (10)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (5) | 5 (15)
Headache (Nervous system disorders) | 2 (3) | 1 (2) | 6 (16)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (4)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 1 (1) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 4 (5)
Insomnia (Psychiatric disorders) | 1 (3) | 0 (0) | 5 (22)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (6)
Proteinuria (Renal and urinary disorders) | 5 (20) | 2 (4) | 24 (84)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (10)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 2 (2) | 7 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (6) | 8 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (10) | 3 (4) | 22 (86)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 4 (6)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 5 (12)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 1 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (9)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (10)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (7) | 7 (9)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (22) | 3 (8) | 13 (43)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (5)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 2 (3)
Hemorrhage (Vascular disorders) | 1 (7) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (9) | 2 (3) | 15 (75)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less